CLINICAL TRIAL: NCT00487448
Title: FLAG-IDA Chemotherapy Induction Follow by Intensive Chemotherapy Postremission +/- Autologous Hemopoietic Stem Cell Transplantation or Bone Marrow Transplantation in Patients With High Risk Myelodysplastic Syndromes or Secondary Acute Myeloblastic Leukemia.
Brief Title: SMD_FLAG-IDA_98: FLAG-IDA in Induction Treatment of High Risk Myelodysplastic Syndromes or Secondary Acute Myeloblastic Leukemia
Acronym: FLAG-IDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Dr Josep Mª Ribera. Executive Secretary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMD_FLAG-IDA_98
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloblastic Leukemia
Keywords: Myelodysplastic Syndrome; Chemotherapy; Peripheral blood stem cells transplantation; Bone marrow transplantation; Secondary Acute Myeloblastic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine; Granulocyte Colony-Stimulating Factor; Idarubicin; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fludarabine
Drug: Cytarabine
Drug: G-CSF
Drug: Idarubicin
Procedure: Peripheral blood stem cell transplantation
Procedure: Bone marrow transplantation

SUMMARY:
Association group of therapeutic specialities authorized in a remission induction treatment(FLAG-IDA: fludarabine, cytarabine, G-CSF (lenograstim) and idarubicin) and an intensive postremission treatment with authorized therapeutic association specialities and with/without Autologous Hemopoietic Stem Cell Transplantation or Bone Marrow Transplantation in Patients With High Risk Myelodysplastic Syndromes or Secondary Acute Myeloblastic Leukemia.

DETAILED DESCRIPTION:
To reach the first remission, the patients receive one cycle of FLAG-IDA combination, that include: Fludarabine 30 mg/m 2 /d Days 1 to 4 in IV perfusion during 30 minutes; Cytarabine 2 g/m 2/d, days 1 to 4 in IV perfusion during 4 hours glycosylate G-CSF 300 µg/m 2/d, days -1 to 5 SC; lenograstim 263 µg/d f, days 11 until absolute neutrophil count >1x10 9 /L SC; Idarubicin 10 mg/m2/d, days 1 to 3 IV bolus (15 minutes)

Patients who don't reach complete remission (CR) are considered as a failure and must go out of study.

The participating centres should decide if the patients under 35 years in CR and with unrelated donor, are excluded to be treated with allogenic transplantation or they continue in the study.

The patients who reach CR will receive one consolidation cycle with IDA-ARAC + G-CSF combination:

Idarubicin 10 mg/m2/d, days 1 to 3 IV bolus (15 minutes); Cytarabine 200 mg/m 2/d days 1 to 5 IV in 24 hours continuous perfusion; glycosylate G-CSF(lenograstim) 263 µg, days 12 until absolute neutrophil count >1x10 9 /L SC

The patients younger than 65 years that is possible, will done an autologous transplantation with peripheral stem blood cells or combined with peripheral stem blood cells and bone marrow stem cells. The preparative regimen recommended are BuCy2 (busulfan-cyclophosphamide) and ICT-Cy (irradiation corporal total-cyclophosphamide).

The patients older than 65 years will receive one intensification cycle with carboplatin and G-CSF.

The peripheral blood stem cells collection should be done during the recuperation period after consolidation chemotherapy in patients under 65 years. The leucapheresis procedure could be determinate for in each center participating.

The patients with no sufficient collection of stem cells during the regeneration period post-chemotherapy of consolidation, will receive glycosylate G-CSF (lenograstim, Granocyte®)10 µg/kg/d SC during 5 days, doing the collection cells on days 5 and 6. In the situations that the peripheral blood stem cells are non satisfactory, will realize a collection of bone marrow stem cells.

The realization of Peripheral Blood Stem Cell Transplantation or combined, depends the number of cells obtained in the collection procedures.In the situations that didn't reach sufficient number of cells (peripheral blood and bone marrow), should be administered one chemotherapy intensification cycle.

The preparative regimen is established by each participating center, but is recommended one of next:

1. BuCy2 (busulfan 16 mg/kg follow by cyclophosphamide 120 mg/kg),
2. Total-body irradiation 12 Gy and cyclophosphamide 120 mg/kg.

Intensification treatment:

Patients older than 65 years and younger than 65 who the collection cells for transplantation is not enough, will receive one cycle of intensification chemotherapy with carboplatin and glycosylate G-CSF:

Carboplatin 300 mg/m2/d days 1 to 4 IV in 24 hours continuous perfusion glycosylate G-CSF (lenograstim)263 µg f days 11 until absolute neutrophil count >1x10 9 /L, SC

ELIGIBILITY:
Inclusion Criteria:

* Age < 75 years
* Diagnosis of Myelodysplastic Syndrome in order to FAB criteria, excluding patients with chronic myeloid leukemia.
* IPI > 1 (High risk or Intermedia risk-2) and/or IPE equal or > 3 (High risk o Intermedia risk) or secondary acute myeloid leukemia.
* Resolved toxicity for previous treatments received to Myelodysplastic Syndrome .
* Myelodysplastic Syndrome de novo.

Exclusion Criteria:

* Associated neoplasia.
* Chronic disease that can limit the patient follow up protocol (cardiovascular disease, active infection uncontrolled, etc.).
* Age < 55 years with related donor HLA compatible.
* Use an investigational drug in the 30 previous days.
* Previous treatment with chemotherapy agents.
* Simultaneous treatment during the study with other drugs not allowed in the protocol.
* Bilirubin > 2 mg/dL and GPT >2 times the normal value.
* Creatinine > 2 mg/dL.
* Hypersensibility to agents used in the protocol.
* Secondary MDS to chemo-radiotherapy .
* HIV positive.
* Chronic myeloblastic leukemia

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1998-07; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of study treatment: complete remission rate, remission duration and global survival | 2 years

SECONDARY OUTCOMES:
Evaluation of neutropenia and thrombocytopenia duration post-induction chemotherapy | 3 months
Determinate the percentage of patients that reach the transplantation | 3 months
Determinate the toxicity of induction regimen and the chemotherapy postremission | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Guillermo, Dr, Study Chair — Hospital La Fe; Sanz Miguel Angel, Dr, Principal Investigator — Hospital La Fe
Locations (15):
- Spain (15):
  - Hospital de la Ribera, Alzira
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital del SAS, Jerez de la Frontera
  - Hospital de Leon, León
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Morales Messeguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Dr. Pesset, Valencia
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org